CLINICAL TRIAL: NCT01796197
Title: Phase II Trial of Paclitaxel Combined With Trastuzumab and Pertuzumab as Pre-Operative Therapy for Inflammatory Breast Cancer
Brief Title: Paclitaxel + Trastuzumab + Pertuzumab as Pre-Op for Inflammatory BrCa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Filipa Lynce, MD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-497
Record Dates: First submitted 2013-02-20; First posted 2013-02-21 (Estimated); Results first posted 2021-09-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Paclitaxel; Doxorubicin; Cyclophosphamide; Mastectomy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Run in: Trastuzumab IV 4 mg/kg, Pertuzumab IV 840 mg (Day 1 Week 1)
  Pre-Op:
  Trastuzumab IV 2 mg/kg weekly, Paclitaxel 80 mg/m2 IV weekly (beginning on Day 8 Week 2) x 16 doses.
  Starting Day 21 (week 4) continue trastuzumab and paclitaxel as above, add Pertuzumab 420 mg IV x 3 weeks. After completing 16 doses of Paclitaxel, Trastuzumab (6 mg/kg IV) and Pertuzumab 420 mg IV may be continued x 3 weeks until surgery Modified Radical Mastectomy
  Post-Op:
  Option 1: Adriamycin 60 mg/m2 IV and Cyclophosphamide 600 mg/m2 IV x 2-3 weeks x 4 cycles. Followed by Trastuzumab 8 mg/kg and Pertuzumab 840 IV load; followed by Trastuzumab 6 mg/kg every and Pertuzumab 420 mg IV every 3 weeks to complete 12 months of HER2-directed therapy Option 2: Continue Trastuzumab 6 mg/kg and Pertuzumab 420 mg x 3 weeks to complete 12 months of HER2-directed therapy Post-mastectomy radiation to the chest wall / regional lymph nodes and endocrine therapy by standard of care.
  Interventions: Drug: Trastuzumab; Drug: Pertuzumab; Drug: Paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Procedure: Mastectomy; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Trastuzumab
Drug: Pertuzumab
Drug: Paclitaxel
Drug: Doxorubicin
Drug: Cyclophosphamide
Procedure: Mastectomy
Radiation: Radiation Therapy

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. In this study, paclitaxel and trastuzumab are being combined with pertuzumab which is "investigational" for the preoperative treatment of inflammatory breast cancer. Trastuzumab is given for a total of 12 months for the treatment of HER2 positive breast cancer. This study also adds pertuzumab to trastuzumab so that both drugs are given for a total of 12 months; this combination is also "investigational".

"Investigational" means that pertuzumab is being studied. It also means that although the FDA has approved pertuzumab for preoperative use to treat breast cancer, it has not been thoroughly studied in combination with paclitaxel and trastuzumab for preoperative treatment of inflammatory breast cancer. It has been FDA approved for specific use in advanced breast cancer that is HER2 positive.

Pertuzumab is an antibody, which is a protein that attacks a foreign substance is the body. Pertuzumab blocks the function of the HER2 protein like trastuzumab does. However, pertuzumab binds to a different part of the HER2 receptor and stops cancer cells from growing. This drug has been used in the treatment of advanced breast cancer that is HER2 positive, and has been combined with trastuzumab and chemotherapy in those studies. Information from those other research studies suggests that pertuzumab may help to kill the cancer cells in the breast and enable you to undergo a mastectomy. The addition of pertuzumab may also help reduce the chance of cancer recurrence.

In this research study, we are combining pertuzumab with paclitaxel and trastuzumab as preoperative therapy and will determine the response of the cancer remaining in the breast at the time of mastectomy. In addition, we are combining trastuzumab with pertuzumab for a total of 12 months and we are looking to see whether the combination reduces the chance that the cancer will return.

Another goal of this research study is to determine whether we can develop a way to identify tumors that will respond well to this study treatment. We will do research tests on your tumor tissue before, during and after study treatment. These tests may help doctors understand how the study treatment may work to treat your type of breast cancer. In the future, these tests may help us find ways to help match patients with the drugs most likely to work against their specific tumors before treatment begins.

DETAILED DESCRIPTION:
If you agree to take part in this study we will ask you to undergo some screening tests and procedures to confirm that you are eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. The screening process will include the following: a medical history, performance status, physical examination, scans and x-rays, blood samples, blood pregnancy test, electrocardiogram, echocardiogram. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria you will not be able to participate in this research study.

Before beginning study treatment you will undergo a tumor biopsy and have photographs of your tumor taken to assess the response of your tumor to the study treatment.

On the first day of study treatment (Week 1, Day 1) with trastuzumab and pertuzumab, you will receive an intravenous infusion of trastuzumab over about 90 minutes, followed by a 60 minutes observation period. If the trastuzumab infusion is tolerated, you will receive the rest of your study treatment, the pertuzumab. This will also be given as an intravenous infusion over about 60 minutes with you being observed for a further 60 minutes. Thus, the total duration of infusion and observation periods for the first dose of study treatment (Week 1, Day 1) is about 5 hours. If the drugs are well tolerated at Week 1, the duration of the infusion with trastuzumab and pertuzumab may be shortened for subsequent doses.

Prior to starting Week 2, you will undergo a second research biopsy of your breast. The biopsy will be performed either prior to Week 2, Day 8 or on the same day. You will then receive an infusion of trastuzumab and begin chemotherapy. If the infusion of trastuzumab was tolerated on Week 1, Day 1, then the infusion time is reduced to about 30 minutes. You will then be pre-medicated with drugs to reduce the chance of having a sensitivity reaction to paclitaxel. This takes approximately 30 minutes. The paclitaxel is give by intravenous infusion over about 60 minutes. If you tolerate the paclitaxel infusions, then the pre-medication can be changed by your doctor.

The pertuzumab is given every 3 weeks beginning on Week 1 and continues until paclitaxel administration is complete. Trastuzumab is given weekly beginning on Week 1 and continues until paclitaxel administration is complete. Paclitaxel is given weekly for a total of 16 doses beginning on Week 2. After completing 16 doses of paclitaxel, trastuzumab and pertuzumab may be continued every 3 weeks until surgery.

Study treatment visits will occur at regular intervals during the period of study treatment, beginning on Week 1. During these study treatment visits the following will be done: physical exam, performance status, blood samples, heart function tests.

After completing 16 doses of paclitaxel in combination with pertuzumab and trastuzumab, you will undergo surgery for removal of your breast cancer. This will occur approximately 4-5 weeks after your last paclitaxel infusion. Prior to surgery, you will have the following assessments: a repeat breast MRI, PET scan (if necessary), physical exam, vital signs, performance status, blood tests, tumor tissue tests.

Approximately 4-5 weeks after surgery, when you are well-healed, you will have two options for treatment (at your physician's discretion):

Option 1: Doxorubicin and cyclophosphamide (AC), every 2-3 weeks x 4 cycles. This is standard chemotherapy for IBC. Followed by trastuzumab and pertuzumab every 3 weeks to complete 12 months of HER2-directed therapy.

Option 2: Continue trastuzumab and pertuzumab every 3 weeks to complete 12 months of HER2-directed therapy.

Doxorubicin is given by vein over about 5-10 minutes. This is followed by cyclophosphamide by vein given about 30 minutes. Anti-nausea medicine is given first under the direction of your doctor.

Approximately 4-5 weeks after finishing the AC treatment if you pursue Option 1 (or 4-5 weeks after surgery if you pursue Option 2), you will receive radiation therapy to the mastectomy site and the surrounding lymph nodes. This will be given daily, Monday through Friday for approximately 6-7 weeks. This will be administered as standard of care for IBC.

Approximately 3-4 weeks following the completion of AC if you pursue Option 1 (or 3-4 weeks after surgery if you pursue Option 2), you will begin maintenance therapy with trastuzumab and pertuzumab. As with Week 1, Day 1, you will receive an intravenous infusion of trastuzumab over about 90 minutes followed by a 60 minute observation period. If the trastuzumab infusion is tolerated, you will receive the rest of your study treatment, the pertuzumab. This will also be given as an intravenous infusion over about 60 minutes with your being observed for a further 60 minutes. Thus, the total duration of infusion and observation periods for the first day of maintenance study treatment is about 5 hours. If the study drugs are well tolerated, the duration of the infusion with trastuzumab and pertuzumab may be shortened for subsequent doses. Both trastuzumab and pertuzumab will be given every 3 weeks to complete a 12 month duration of HER2-directed therapy. Every 9 weeks (every third dose of trastuzumab and pertuzumab) you will undergo the same procedure as taht described above in Study Treatment visits.

About one month after your last dose of study treatment, you will be asked to return to the clinic. At this visit tests will be done to check your physical condition and to check that you have recovered from any side effects of study treatment. During this visit the following will be done: physical exam, vital signs, performance status and blood tests.

You will be asked to attend regular follow up visits to check if you are experiencing any long term side effects and to check taht the cancer has not come back. We plan to follow participants for up to 13 years after the start of teh study. During these visits the following will be done: physical exam and questions about your health/medications you have taken (every 3 months for the first year, every 6 months for the next 4 years, yearly until the end of study follow up); blood draws (every 6 months for the first 4 years, yearly after that); mammograms will be performed annually, other scans may be performed as needed.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer
* HER2 positive breast cancer
* Clinical diagnosis of inflammatory breast cancer
* Without evidence of visceral or bone involvement with metastatic cancer on physical exam or any diagnostic study. Extensive nodal involvement is allowed
* Willingness to undergo a research biopsy of the affected breast

Exclusion Criteria:

* Prior therapy for the treatment of breast cancer
* Receiving any other investigational or commercial agents or therapies
* Known brain metastases
* Symptomatic intrinsic lung disease or extensive tumor involvement of the lungs resulting in dyspnea at rest
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to paclitaxel, trastuzumab, pertuzumab
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding
* History of a different malignancy except for the following circumstances: disease-free for at least 5 years and at low risk of recurrence, or cervical cancer in situ or basal or squamous cell carcinoma of the skin
* HIV positive on combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2026-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Filipa Lynce, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan

REFERENCES:
- [Derived] Pernas S, Guerriero JL, Naumenko S, Goel S, Regan MM, Hu J, Harrison BT, Lynce F, Lin NU, Partridge A, Morikawa A, Hutchinson J, Mittendorf EA, Sokolov A, Overmoyer B. Early on-treatment transcriptional profiling as a tool for improving pathological response prediction in HER2-positive inflammatory breast cancer. Ther Adv Med Oncol. 2022 Jul 30;14:17588359221113269. doi: 10.1177/17588359221113269. eCollection 2022. PMID 35923923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: August 2013 to June 2018
Pre-assignment Details: Participants are not being evaluated based on their post-operative treatment option. Two options are provided to the participants in order to best treat them based on the nature of their disease.
Groups:
- Treatment Arm: Run in phase: Trastuzumab IV 4 mg/kg, Pertuzumab IV 840 mg (Day 1, Week 1)
  Pre-op phase:
  Trastuzumab IV 2 mg/kg weekly, Paclitaxel 80 mg/m2 IV weekly (beginning on Day 8, Week 2) x 16 doses.
  Starting Day 21 (week 4) continue trastuzumab and paclitaxel as above and add Pertuzumab 420 mg IV every 3 weeks during 16 doses of paclitaxel administration. After completing 16 doses of Paclitaxel, Trastuzumab (6 mg/kg IV) and Pertuzumab 420 mg IV may be continued every 3 weeks until surgery
  Modified Radical Mastectomy
  Post-Operative Treatment (Two Options):
  Option 1: Adriamycin 60 mg/m2 IV and Cyclophosphamide 600 mg/m2 IV every 2-3 weeks x 4 cycles. Followed by Trastuzumab 8 mg/kg and Pertuzumab 840 IV load; followed by Trastuzumab 6 mg/kg every and Pertuzumab 420 mg IV every 3 weeks to complete 12 months of HER2-directed therapy
  Option 2: Continue Trastuzumab 6 mg/kg and Pertuzumab 420 mg every 3 weeks to complete 12 months of HER2-directed therapy
  Post-mastectomy radiation therapy to the chest wall and regional lymph nodes and endocrine therapy administered to participants by standard of care.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 23
Completed | 21
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Participants are not being evaluated based on their post-operative treatment option. Two options are provided to the participants in order to best treat them based on the nature of their disease
Arm/Group | Treatment Arm
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 48 [32 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 23
Estrogen Receptor Status [Count of Participants; unit: Participants]
  Negative | 11
  Positive | 12
Breast Cancer Stage [Count of Participants; unit: Participants] — IIIB:
  Tumor may be any size and has spread to the chest wall and/or skin of the breast and caused swelling or an ulcer and may have spread to >10 axillary lymph nodes or spread to lymph nodes near breastbone.
  IIIC:
  May be no sign of cancer in the breast or, tumor may be any size and may have spread to the chest wall and/or the skin of the breast and 10 or more axillary lymph nodes or lymph nodes above or below the collarbone or spread to axillary lymph nodes or to lymph nodes near the breastbone
  IV:
  Spready beyond the breast and nearby lymph nodes.
  Participants
    IIIB | 16
    IIIC | 6
    IV | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Participants With Pathologic Complete Response
Description: Pathologic complete response (pCR) is defined as absence of invasive carcinoma within the breast and axillary lymph nodes following preoperative treatment. Participants whose disease is not surgically resectable following preoperative treatment are considered as not having pCR.
Time Frame: 18 weeks
Population: Subjects evaluable for response. Participants are not being evaluated based on their post-operative treatment option. Two options are provided to the participants in order to best treat them based on the nature of their disease
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
percentage of participants | 48 [29 to 67]
Statistical Analysis 1: Comparison: Treatment Arm; Null Hypothesis: pCR rate is less than or equal to 15% Alternative Hypothesis: pCR rate is greater than or equal to 40% Hypothesized False Positive Rate (alpha) : 3.9% Hypothesized False Negative Rate (1-beta) : 9.9%; Test type: Superiority; Two stage design, exact method; Pathelogic Complete Response Rate = 40 — Decision Rule: If the percentage of participants experiencing pathologic complete response (pCR) is ≤ 15% then the preoperative regimen is considered minimally effective. If the proportion of pCR ≥ 40% then the regimen is worthy of further study

2. Primary Outcome: Residual Cancer Burden Rate
Description: Residual cancer burden is calculated an then categorized based on the methods described in the following: Symmans WF, Peintinger F, Hatzis C, et al. Measurement of residual breast cancer burden to predict survival after neoadjuvant chemotherapy. J Clin Oncol 2007;25(28): 4414-22.
  This method uses tumor size, the proportion of that tumor that is invasive carcinoma, the number of axillary lymph nodes containing metastatic carcinoma and the diameter of the largest metastasis in an axillary lymph node. These parameters are combined in a formula that outputs a RCB index. This index is divided into 4 categories: RCB-0, RCB-I, RCB-II, and RCB-III. The previous categories are in order of increasing severity of RCB.
Time Frame: 18 Weeks
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
percentage of participants
  RCB-0 | 48 [29 to 67]
  RCB-I | 33 [17 to 54]
  RCB-II | 5 [2 to 21]
  RCB-III | 14 [4 to 33]

3. Secondary Outcome: Number of Participants With Congestive Heart Failure
Description: Number of participants with clinically significant congestive heart failure (CHF) as determined by established medical practices.
Time Frame: 1 year and 8 months
Population: Participants evaluable for adverse events. Participants are not being evaluated based on their post-operative treatment option. Two options are provided to the participants in order to best treat them based on the nature of their disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 23
Participants | 0

4. Secondary Outcome: Median Disease Free Survival
Description: Disease-free survival (DFS) is defined for the participants who undergo surgery, as the duration of time from surgery until ipsilateral local-regional, contralateral or distant invasive recurrence or death from any cause; in the absence of an event, DFS will be censored at the date last know alive and free from recurrence.
Time Frame: 63 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
months | NA [NA to NA] — Less than 50% recurrence at the time of data extraction, so median DFS not reached. It is not possible to calculate the lower limit of the confidence interval.

5. Secondary Outcome: Median Time to Treatment Failure
Description: Time to treatment failure (TTF) will be defined among all participants, as the duration of time from treatment initiation to a DFS event or progressive disease during preoperative therapy or treatment disease that is not surgically resectable; in the absence of an event, TTF will be censored at the date last know alive and free from recurrence or progression.
Time Frame: 63 months
Population: Subjects evaluable for response. Two options are provided to the participants in order to best treat them based on the nature of their disease.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
months | NA [NA to NA] — Less than 50% recurrence at the time of data extraction, so median TTF not reached. Participants are not being evaluated based on their post-operative treatment option. It is not possible to calculate the lower limit of the confidence interval.

6. Secondary Outcome: Median Overall Survival
Description: Overall survival (OS) will be defined among all participants, as the duration of time from treatment initiation to death from any cause, or is censored at date last known alive. Post-surgery OS will be defined among the participants who undergo surgery, as the duration of time from treatment initiation to death from any cause, or is censored at date last known alive.
Time Frame: 63 months
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
months | NA [NA to NA] — Less than 50% recurrence at the time of data extraction, so median OS not reached. Participants are not being evaluated based on their post-operative treatment option. It is not possible to calculate the lower limit of the confidence interval.

7. Secondary Outcome: Pathological Complete Response Rate by Intrinsic Subtype
Description: Pathologic complete response (pCR) is defined as absence of invasive carcinoma within the breast and axillary lymph nodes following preoperative treatment. Participants whose disease is not surgically resectable following preoperative treatment are considered as not having pCR. PAM50 analysis was performed on the biopsy specimen taken on day 1.
  Participants' pCR was tabulated according to the intrinsic subtype and the association of intrinsic subtype (Estrogen receptor 2 - enriched vs. other) with pCR was assessed using Fisher's exact test.
Time Frame: 18 Weeks
Population: No samples collected since very few patients had residual disease and sample size would be too small for any meaningful analysis.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

8. Secondary Outcome: Residual Disease Rate by Intrinsic Subtype
Description: Residual Disease Rate is the percentage of participants who do not achieve Pathologic complete response (pCR) by the end of preoperative treatment. pCR is defined as absence of invasive carcinoma within the breast and axillary lymph nodes following preoperative treatment. Residual disease within the breast at time of mastectomy was assessed by microarray analysis. Residual disease rate was reported by intrinsic subtype identified using day 1 RNAseq analysis.
Time Frame: 18 Weeks
Population: as for outcome 7
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

9. Secondary Outcome: Predictive Accuracy Rate of Pre-Treatment Versus On-Treatment Tumor Biopsy RNA Sequencing Profiles
Description: Tumor RNA expression from pre-treatment (Day 1) and on-treatment (Day 8) biopsies were evaluated to see if the expression profiles had predictive accuracy of pCR. pCR is defined as absence of invasive carcinoma within the breast and axillary lymph nodes following preoperative treatment. Participants whose disease is not surgically resectable following preoperative treatment are considered as not having pCR. The biopsies were analyzed by differential expression analysis using standard procedures in R package, limma. A predictive Random Forest model was trained using leave-pair-out-cross-validation with the 80 genes most associated with pCR and/or non-pCR. This model gives an accuracy rate, which indicates the percentage of time that the gene profile predicts pCR or non-pCR for both the pre-treatment and on-treatment profiles. An increase in accuracy for the on-treatment profile would indicate an adaptive response within the tumor associated with resistance to HER2 directed therapies.
Time Frame: 18 Weeks
Population: as for outcome 5
Measure: Number; unit: percent accuracy
Arm/Group | Treatment Arm
Number analyzed (Participants) | 21
percent accuracy
  Day 1 Biopsy | 50
  Day 8 Biopsy | 90

10. Secondary Outcome: Residual Cancer Burden Rate by ctDNA Profile Change
Description: Residual cancer burden is calculated an then categorized based on the methods described in the following: Symmans WF, Peintinger F, Hatzis C, et al. Measurement of residual breast cancer burden to predict survival after neoadjuvant chemotherapy. J Clin Oncol 2007;25(28): 4414-22.
  This method uses tumor size, the proportion of that tumor that is invasive carcinoma, the number of axillary lymph nodes containing metastatic carcinoma and the diameter of the largest metastasis in an axillary lymph node. These parameters are combined in a formula that outputs a RCB index. This index is divided into 4 categories: RCB-0, RCB-I, RCB-II, and RCB-III. The previous categories are in order of increasing severity of RCB.
  Biopsy/blood will be collected on day 1 and day 8 of therapy for analysis of circulating biomarkers, including ctDNA.
  Associations between change in ctDNA during therapy and residual cancer burden at the time of definitive surgery will be evaluated.
Time Frame: 18 weeks
Population: Data was not collected due to a lack of clinical research funding.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 63 Months
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. Remaining AEs are classified as Other AEs (OAE). Maximum grade toxicity by type was calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term. Participants are not being evaluated based on their post-operative treatment option.
Groups:
- Treatment Arm: Pre-op phase:
  Trastuzumab: IV 4mg/kg/first dose, then IV 2mg/kg weekly. Pertuzumab: IV 840mg/first dose, then IV 420mg every 3 weeks Paclitaxel: IV 80mg/m2 weekly x 16 doses Trastuzumab (6 mg/kg IV) and Pertuzumab 420 mg IV may be continued every 3 weeks until surgery.
  Surgery: Modified Radical Mastectomy
  Post-Operative Treatment:
  Option 1: Adriamycin 60 mg/m2 IV and Cyclophosphamide 600 mg/m2 IV every 2-3 weeks x 4 cycles. Followed by Trastuzumab 8 mg/kg and Pertuzumab 840 IV load; followed by Trastuzumab 6 mg/kg every and Pertuzumab 420 mg IV every 3 weeks to complete 12 months of HER2-directed therapy
  Option 2: Continue Trastuzumab 6 mg/kg and Pertuzumab 420 mg every 3 weeks to complete 12 months of HER2-directed therapy
  All patients should also complete radiation therapy.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 6/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Alkaline phosphatase increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=23)
Anemia (Blood and lymphatic system disorders) | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Lymph node pain (Blood and lymphatic system disorders) | 3
Ear pain (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Blurred vision (Eye disorders) | 4
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Cheilitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 19
Dry mouth (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 10
Nausea (Gastrointestinal disorders) | 11
Rectal hemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Edema limbs (General disorders and administration site conditions) | 3
Edema trunk (General disorders and administration site conditions) | 1
Fatigue (General disorders and administration site conditions) | 20
Fever (General disorders and administration site conditions) | 2
Flu like symptoms (General disorders and administration site conditions) | 2
Gait disturbance (General disorders and administration site conditions) | 2
Infusion related reaction (General disorders and administration site conditions) | 5
Localized edema (General disorders and administration site conditions) | 2
Non-cardiac chest pain (General disorders and administration site conditions) | 1
Pain (General disorders and administration site conditions) | 3
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Eye infection (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Infections and infestations - Other, specify (Infections and infestations) | 3
Dermatitis radiation (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 3
Creatinine increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Growth suppression (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Cognitive disturbance (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 7
Extrapyramidal disorder (Nervous system disorders) | 1
Facial muscle weakness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 7
Movements involuntary (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 15
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 6
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 3
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Vaginal inflammation (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 3
Nail loss (Skin and subcutaneous tissue disorders) | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 3
Periorbital edema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6
Hot flashes (Vascular disorders) | 4
Lymphedema (Vascular disorders) | 3
Thromboembolic event (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-23): https://cdn.clinicaltrials.gov/large-docs/97/NCT01796197/Prot_SAP_000.pdf